CLINICAL TRIAL: NCT07124182
Title: Chewing Gum During a Pap Smear: A Randomized Controlled Clinical Trial
Brief Title: Chewing Gum During a Pap Smear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, NURDİLAN SENER, Head of the Department of Obstetrics and Gynecology Nursing, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: fıratuniverstyyy; fırat unversity (Other: fırat universty)
Record Dates: First submitted 2025-08-03; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Woman Aged 18 to 65; Woman of Reproductive Age
Keywords: pap smear; pain; anxiety; gum
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled trial was conducted to determine the effects of chewing gum on anxiety and pain in women during pap smears.
Who Masked: Participant
Masking Description: Block randomization was used to assign participants to the experimental and control groups to ensure equal distribution between groups. Block randomization reduced selection bias and ensured uniformity in group size. A block size of four was set at four, ensuring that two participants were assigned to the intervention group and two to the control group. Using SPSS 25.0 statistical software, all possible group combinations (e.g., DDKK, KDKD, DKDK, KKDD, etc.) were randomly generated to achieve a 1:1 assignment ratio. Group assignments within each combination were placed individually in envelopes with envelope numbers, the contents of which were hidden from view. Participants were asked to randomly select one of these envelopes in the order they arrived at the clinic before data collection. Participants were assigned to the relevant group based on the group information written inside the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (chewing gum) (Experimental): Participants in the experimental group were given gum after the pretest and asked to chew it. They were asked to chew it until they stepped off the gynecological examination table. The women chewed gum for an average of 10 minutes. The gum they were given was unflavored and sugar-free.
  Interventions: Other: shewing gum
- control group (no intervention) (No Intervention): Participants in the control group received no intervention.

INTERVENTIONS:
Other: shewing gum — Chewing gum is a cost-effective practice that can provide comfort to women. A Pap smear is an important test. Women experiencing pain, anxiety, or other symptoms may discourage testing. Chewing gum can reduce these sensitivities.
  Arms: experimental group (chewing gum)

SUMMARY:
This study, which was conducted to determine the effects of chewing gum on anxiety and pain during Pap smear, found that chewing gum reduced pain but had no effect on anxiety.

DETAILED DESCRIPTION:
Cervical cancer is one of the most common malignancies in women aged 35-44. Cervical cancer screening methods include the Papanicolaou test (PAP) via cytopathology, and the Pap smear is widely used for early detection of cervical cancer. A Pap smear involves a speculum examination, direct visualization of the cervix, and collection of a sample from the cervix using a brush. ACOG recommends screening for women aged 30-65 with cervical cytology alone every 3 years, with high-risk HPV testing alone every 5 years, or with cytology and high-risk HPV testing (concurrent testing) every 5 years (ACOG).

Women often experience anxiety and pain during pelvic procedures. Anxiety is a distressing emotional state. Many women with increased anxiety are at risk of experiencing pain. An adrenergic response is activated between the physiological effects of anxiety and the perception of pain. It has been reported that the pap smear procedure, which is a pelvic procedure, is relatively short, and cognitive and behavioral interventions that distract the patient can be effective in reducing pain and anxiety. In addition, strategies for alleviating pain and anxiety include pharmacological and non-pharmacological interventions. Non-pharmacological methods are reported to be inexpensive and easy to implement, and have relatively few side effects. Various interventions, such as booklets, brochures, informative videos, education, and music, have been tested in the literature to reduce anxiety and pain levels. Neuropsychology confirms that chewing gum increases sustained attention. Chewing gum has a sustained effect on alertness and attention. Chewing gum can lower cortisol levels, reduce distractions, and increase cognitive focus. This can reduce overall stress and anxiety. Chewing gum is reported to be a cheap, well-tolerated, safe, and effective way to alleviate anxiety and stress . There are no direct studies in the literature on the use of gum during Pap smears. This study aimed to examine the effect of chewing gum during Pap smears.

ELIGIBILITY:
Inclusion Criteria:

* Women who are literate, can speak and understand Turkish, are not pregnant, are not in menopause, and have experienced sexuality

Exclusion Criteria:

* women diagnosed with cervical cancer

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pap smear with vaginal examination is only suitable for women
Enrollment: 103 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in pain level during Pap smear procedure | Immediately after completion of the Pap smear procedure (within approximately 10 minutes)
  Change from baseline in self-reported pain score, measured using the Visual Analog Scale (VAS; 0-10), during and immediately after the Pap smear procedure
Change in anxiety level during gynecological examination | Immediately after completion of the gynecological examination (within approximately 10 minutes)
  Change from baseline in self-reported anxiety score, measured using the State-Trait Anxiety Inventory (STAI; range 20-80), during and immediately after the gynecological examination

CONTACTS AND LOCATIONS:
Locations (1):
- Firat Universty, Elâzığ, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No